CLINICAL TRIAL: NCT03282097
Title: Decisions About Cancer Screening in Alzheimer's Disease
Acronym: DECAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1501278953; 5R01AG055424 (NIH)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer, Breast; Alzheimer Disease
MeSH Terms: conditions — Breast Neoplasms; Alzheimer Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mammogram decision aid (Experimental): Family caregivers and patients with dementia will be mailed the DECAD decision aid about mammography and breast cancer screening before the patients next PCP visit to test if the aid improves decision making about breast cancer screening in older women with dementia.
  Interventions: Behavioral: DECAD decision aid
- Home safety guide (Active Comparator): Family caregivers and patients with dementia will be mailed a home safety guide, which is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group about mammography.
  Interventions: Other: Home safety guide

INTERVENTIONS:
Behavioral: DECAD decision aid — A mammography decision aid directed toward family caregivers of older women with Alzheimer's disease and other dementias to assist with decisions about breast cancer screening.
  Arms: Mammogram decision aid
Other: Home safety guide — The home safety guide to provide tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
  Other Names: control group
  Arms: Home safety guide

SUMMARY:
The Decisions about Cancer screening in Alzheimer's Disease (DECAD) study tests if an evidence-based decision aid for dementia caregivers can support decision-making about mammography and improve the quality of medical decision-making about breast cancer screening. This large randomized controlled trial will recruit up to 450 dyads (900 individual participants) of older women with dementia and a family caregiver, for a goal of 426 dyad baselines (852 individual participants).

DETAILED DESCRIPTION:
Alzheimer's disease and related dementias (ADRD) impact a woman's life expectancy and her ability to participate in medical decision-making about breast cancer screening, necessitating the involvement of family caregivers. Making decisions about mammography screening for women with ADRD is stressful. There are no data that suggest that breast cancer screening helps women with ADRD live longer or better. Decision aids may improve the quality of decision-making about mammography for ADRD patients and may inform family caregivers about the risks, benefits, and need for decision-making around mammography screening.

The Decisions about Cancer Screening in Alzheimer's Disease (DECAD) trial, a randomized controlled clinical trial, will enroll 426 dyads of older women with ADRD (≥75 years) and a family caregiver from clinics and primary-care practices to test a novel, evidence-based decision aid. This decision aid includes information about the impact of ADRD on life expectancy, the benefit of mammograms, and the impact on the quality of life for older women with ADRD. Dyads will be randomized to receive the decision aid or active control information about home safety. This trial will examine the effect on the caregiver's decisional conflict (primary outcome) and the caregiver's decision-making self-efficacy (secondary outcome). A second follow-up at 15 months will include a brief, semi-structured interview with the caregiver regarding the patient's experience with mammograms and decision-making about mammograms. At the same time, a review of the patient's electronic medical record (EMR) will look at discussions about mammography with their primary-care physician and mammogram orders, receipt, results, and burden (e.g., additional diagnostic procedures due to false-positive results, identification of an abnormality on the screening exam but further work-up declined, and identification of a clinically unimportant cancer).

We hypothesize that caregivers who receive the decision aid will have lower levels of decisional conflict and higher levels of decision-making self-efficacy compared to the control group. We also hypothesize that the DECAD decision aid will reduce mammography use among older women with ADRD.

ELIGIBILITY:
Patient Inclusion Criteria:

* Female and 75 years or older
* At least one mammogram in the past five years
* Primary care visit scheduled in the next 12 months
* Diagnosis of Alzheimer's disease or related dementia as determined by ICD-10 code
* Ability to provide informed consent or assent
* Ability to communicate in English

Patient Exclusion Criteria:

* Permanent resident of a nursing facility
* Had a mammogram in the past 6 months
* Primary care visit scheduled is the first visit with the PCP
* Made a decision to stop getting mammograms
* History of Atypical Ductal Hyperplasia, lobular carcinoma in situ, ductal carcinoma in situ, or non-invasive breast cancer
* Has mild cognitive impairment, serious mental illness such as bipolar or schizophrenia as determined by ICD-10 code

Caregiver Inclusion Criteria:

* 18 years or older
* Primary family caregiver of the patient*
* Must have a telephone
* Ability to provide informed consent
* Ability to communicate in English

Caregiver Exclusion Criteria:

* Caregiver is a non-family member who is not a legal Healthcare Power of Attorney
* Less than a 7th grade education**
* Made a decision that the patient will stop getting mammograms
* Has a diagnosis of AD or has a serious mental illness such as bipolar or schizophrenia as determined by ICD-10 code

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 442 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fowler, PhD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - Parkview Health, Fort Wayne, Indiana
  - Alzheimer's Association, Indianapolis, Indiana
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fowler NR, Schonberg MA, Sachs GA, Schwartz PH, Gao S, Lane KA, Inger L, Torke AM. Supporting breast cancer screening decisions for caregivers of older women with dementia: study protocol for a randomized controlled trial. Trials. 2018 Dec 12;19(1):678. doi: 10.1186/s13063-018-3039-z. PMID 30541634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from primary care clinics in central Indiana and Boston, MA between November 2017 and August 2022. The first participant was enrolled on December 1, 2017 and the last participant was enrolled on August 29, 2022.
Pre-assignment Details: Of the 442 enrolled dyads, 429 were randomized to receive the mammogram decision aid or home safety pamphlet, 427 dyads met inclusion criteria to proceed with the study.
Groups:
- Mammogram Decision Aid: Will be mailed the DECAD decision aid before their next PCP visit in order to better inform their decision to continue or stop mammography.
  DECAD decision aid: A mammography decision aid that will help caregivers of patients with Alzheimer's make decisions about stopping or continuing breast cancer screening.
- Home Safety Guide: The home safety guide is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group away from talking about mammography with the patient's PCP.
  Home safety guide: The home safety guide provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
Period: Randomized and Completed Baseline
Arm/Group | Mammogram Decision Aid | Home Safety Guide
Started | 214 (This number represents the dyad, both patient and caregiver. There were 214 patients and 214 caregivers enrolled to the Mammogram decision aid arm.) | 215 (This number represents the dyad, both patient and caregiver. There were 215 patients and 215 caregivers enrolled to the Home safety guide arm.)
Completed | 213 (This number represents the dyad, both patient and caregiver. There were 213 patients and 213 caregivers that completed a baseline in the Mammogram decision aid arm.) | 214 (This number represents the dyad, both patient and caregiver. There were 214 patients and 214 caregivers that completed a baseline in the Home safety guide arm.)
Not Completed | 1 | 1
Not completed — Randomized no Baseline | 1 | 1
Period: Intervention Visit Complete
Arm/Group | Mammogram Decision Aid | Home Safety Guide
Started | 213 | 214
Completed | 171 | 155
Not Completed | 42 | 59
Not completed — Patient Death | 13 | 15
Not completed — Caregiver Death | 0 | 3
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Became Ineligible before PCP Index visit | 12 | 21
Not completed — PCP Index Visit Not Completed | 3 | 7
Period: Primary Outcome Data Collection Complete
Arm/Group | Mammogram Decision Aid | Home Safety Guide
Started | 171 | 155
Completed | 168 | 152
Not Completed | 3 | 3
Not completed — Missing | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Period: 15 Month Follow-up Complete
Arm/Group | Mammogram Decision Aid | Home Safety Guide
Started (Dyads that missed the primary outcome data collection visit still had the opportunity to complete 15 month follow up interview.) | 170 | 155
Completed | 164 | 146
Not Completed | 6 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Population: Participant Flow shows the total enrolled dyads (patient and their enrolled caregiver). Baseline Population characteristics reflects both caregiver and patient demographics.
Groups:
- Mammogram Decision Aid - Caregivers; Mammogram Decision Aid - Patient: Will be mailed the DECAD decision aid before their next PCP visit in order to better inform their decision to continue or stop mammography.
  DECAD decision aid: A mammography decision aid that will help caregivers of patients with Alzheimer's make decisions about stopping or continuing breast cancer screening.
- Home Safety Guide - Caregivers; Home Safety Guide - Patient: The home safety guide is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group away from talking about mammography with the patient's PCP.
  Home safety guide: The home safety guide provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
- Total: Total of all reporting groups
Arm/Group | Mammogram Decision Aid - Caregivers | Mammogram Decision Aid - Patient | Home Safety Guide - Caregivers | Home Safety Guide - Patient | Total
Number analyzed (Participants) | 213 | 213 | 214 | 214 | 854
Age, Categorical [Count of Participants; unit: Participants] — Population: 4 participants (caregivers) did not provide age
  Participants
    number analyzed (Participants) | 211 | 213 | 212 | 214 | 850
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 146 | 0 | 139 | 0 | 285
    >=65 years | 65 | 213 | 73 | 214 | 565
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 133 | 213 | 131 | 214 | 691
  Male | 80 | 0 | 82 | 0 | 162
  Other | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 57 | 55 | 51 | 53 | 216
  White | 147 | 150 | 159 | 159 | 615
  Other | 9 | 7 | 4 | 2 | 22
  No response provided | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 213 | 213 | 214 | 214 | 854

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale
Description: The Decisional Conflict Scale (DCS) includes 16-items on a 1-5 Likert scale. Questions are regarding a medical decision that participants have made or that they are about to make; it measures uncertainty around a decision, whether one feels informed, clear about their personal values, and supported in their decision-making It is a validated and widely accepted measure of decision quality that has been used in previous studies of decision aids intended for AD caregivers. Scores can range from 0-100, with lower scores indicating less conflict. This survey is completed during the baseline and Post-Index PCP visit.
Time Frame: Change in DCS score from Baseline to post-PCP Index Visit. Post-PCP Index visit routinely occurs 0-5 days after the patient's index visit with their PCP.
Population: The above values represent the number of dyads that completed the Decisional Conflict Scale (DCS) at both baseline and post-PCP Index Visit.
Measure: Mean (Standard Deviation); unit: Units on DCS scale
Arm/Group | Mammogram Decision Aid | Home Safety Guide
Number analyzed (Participants) | 167 | 152
Units on DCS scale | -1.9 (16.1) | -0.8 (12.0)
Statistical Analysis 1: Comparison: Mammogram Decision Aid vs Home Safety Guide; Test type: Superiority; p = 0.4393, ANCOVA

2. Secondary Outcome: Change in Decision-making Self-efficacy Scale Score
Description: To measure decision-making self-efficacy, we will use the Decision Self-Efficacy Scale (DSE). The DSE is a validated, 11-item instrument that measures how confident the respondent is in their ability to make an informed medical decision, including SDM. We will adapt the DSE with five response categories on a 0-4 Likert scale ("not at all confident", "somewhat confident", "neither confident nor not confident", "confident", and "very confident") to measure caregiver decision-making self-efficacy for mammography decisions for their relative with Alzheimer's Disease and related dementias. To score the sum of all items are divided by 11 and multiplied by 25. Scores range from 0 (Extremely low self-efficacy) to 100 (Extremely high self-efficacy). To measure the change in self-efficacy over time in both groups, we will measure it at two time points.
Time Frame: Change in Decision Self-Efficacy score from Baseline to post-PCP Index Visit. Post-PCP Index visit routinely occurs 0-5 days after the patient's index visit with their PCP.
Population: The above values represent the number of dyads that completed the Decision Self-Efficacy Scale (DSE) at both baseline and post-PCP Index Visit.
Measure: Mean (Standard Deviation); unit: Units on the DSE scale
Groups:
- Mammogram Decision Aid-Family Member: Family caregivers and patients with dementia will be mailed the DECAD decision aid about mammography and breast cancer screening before the patients next PCP visit to test if the aid improves decision making about breast cancer screening in older women with dementia.
  DECAD decision aid: A mammography decision aid directed toward family caregivers of older women with Alzheimer's disease and other dementias to assist with decisions about breast cancer screening.
- Home Safety Guide-Family Member: Family caregivers and patients with dementia will be mailed a home safety guide, which is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group about mammography.
  Home safety guide: The home safety guide to provide tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
Arm/Group | Mammogram Decision Aid-Family Member | Home Safety Guide-Family Member
Number analyzed (Participants) | 167 | 152
Units on the DSE scale | -1.7 (14.6) | 0.0 (11.4)
Statistical Analysis 1: Comparison: Mammogram Decision Aid-Family Member vs Home Safety Guide-Family Member; Test type: Superiority; p = .2262, ANCOVA

3. Secondary Outcome: Caregiver Role in Decision Making
Description: On a scale from 1 to 10, caregivers assessed the role that they have in decision making for the patient. The scale is 1 to 10 where 1 means the patient makes all the medical decisions on her own, 5 means that the patient and caregiver equally share the medical decisions, and 10 means that the caregiver makes all medical decisions for the patient.
Time Frame: The above values represent the number of caregivers that completed the assessment at post-PCP Index Visit. Post-PCP Index visit routinely occurs 0-5 days after the patient's index visit with their PCP.
Population: Caregivers who completed post-PCP Index Visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mammogram Decision Aid-Caregiver: Family caregivers and patients with dementia will be mailed the DECAD decision aid about mammography and breast cancer screening before the patients next PCP visit to test if the aid improves decision making about breast cancer screening in older women with dementia.
  DECAD decision aid: A mammography decision aid directed toward family caregivers of older women with Alzheimer's disease and other dementias to assist with decisions about breast cancer screening.
- Home Safety Guide-Caregiver: Family caregivers and patients with dementia will be mailed a home safety guide, which is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group about mammography.
  Home safety guide: The home safety guide to provide tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
Arm/Group | Mammogram Decision Aid-Caregiver | Home Safety Guide-Caregiver
Number analyzed (Participants) | 168 | 152
units on a scale | 5.7 (1.6) | 5.2 (1.4)
Statistical Analysis 1: Comparison: Mammogram Decision Aid-Caregiver vs Home Safety Guide-Caregiver; Test type: Superiority; p = 0.0023, ANCOVA

4. Secondary Outcome: Receipt of Mammogram Screening
Description: Receipt of mammograms was assessed 15 months post intervention.
Time Frame: 15 month post intervention
Population: All patients who completed an index visit
Measure: Count of Participants; unit: Participants
Groups:
- Mammogram Decision Aid-Patient: Family caregivers and patients with dementia will be mailed the DECAD decision aid about mammography and breast cancer screening before the patients next PCP visit to test if the aid improves decision making about breast cancer screening in older women with dementia.
  DECAD decision aid: A mammography decision aid directed toward family caregivers of older women with Alzheimer's disease and other dementias to assist with decisions about breast cancer screening.
- Home Safety Guide-Patient: Family caregivers and patients with dementia will be mailed a home safety guide, which is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group about mammography.
  Home safety guide: The home safety guide to provide tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
Arm/Group | Mammogram Decision Aid-Patient | Home Safety Guide-Patient
Number analyzed (Participants) | 171 | 155
Participants
  Received mammogram | 32 | 33
  Did not receive mammogram | 139 | 122
Statistical Analysis 1: Comparison: Mammogram Decision Aid-Patient vs Home Safety Guide-Patient; Test type: Superiority; p = 0.6075, Regression, Logistic

5. Secondary Outcome: Change in Caregiver Knowledge About Mammograms in Older Women With ADRD
Description: Knowledge about mammograms for older women with Alzheimer's Disease and Related Dementias will be measured with a 16-item measure (6 multiple choice and 10 true/false) mapped directly from the information presented in the decision aid. Scoring for this study created measure is the sum of the correct responses.
Time Frame: Change in Caregiver knowledge from Baseline to post-PCP Index Visit. Post-PCP Index visit routinely occurs 0-5 days after the patient's index visit with their PCP.
Population: The above values represent the number of caregivers that completed the knowledge assessment at both baseline and post-PCP Index Visit.
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Mammogram Decision Aid-Caregiver | Home Safety Guide-Caregiver
Number analyzed (Participants) | 168 | 152
Units on the scale | 1.4 (2.4) | 0.1 (1.9)
Statistical Analysis 1: Comparison: Mammogram Decision Aid-Caregiver vs Home Safety Guide-Caregiver; Test type: Superiority; p < .0001, ANCOVA

6. Secondary Outcome: Caregiver Intention for the Patient to Receive Mammogram Screening in the Future
Description: Caregivers were asked when they believed the patient would receive their next mammogram. Never responses were labeled as no, and responses that indicated an intention to be screened in the future were labeled as yes.
Time Frame: Post-PCP Index visit routinely occurs 0-5 days after the patient's index visit with their PCP.
Population: The above values represent the number of caregivers that completed the assessment at post-PCP Index Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Mammogram Decision Aid-Caregiver | Home Safety Guide-Caregiver
Number analyzed (Participants) | 159 | 141
Participants
  Yes | 73 | 104
  No | 86 | 37
Statistical Analysis 1: Comparison: Mammogram Decision Aid-Caregiver vs Home Safety Guide-Caregiver; Test type: Superiority; p < 0.0001, Regression, Logistic

ADVERSE EVENTS:
Time Frame: All adverse events, unanticipated problems and potential risks will be monitored and collected ongoing and throughout the study by the DECAD research staff and coordinators. For all patients, adverse events will be collected starting at enrollment and continue until after the patient has completed the study either by completing the 15-month follow up or 24-months post-Primary Outcome Data Collection.
Description: Adverse events or serious adverse events are only collected for the patient in each dyad.
Groups:
- Mammogram Decision Aid - Caregiver: Will be mailed the DECAD decision aid before their next PCP visit in order to better inform their decision to continue or stop mammography.
  DECAD decision aid: A mammography decision aid that will help caregivers of patients with Alzheimer's make decisions about stopping or continuing breast cancer screening.
- Home Safety Guide - Caregiver: The home safety guide is a two-page paper pamphlet developed by the American Geriatrics Society Foundation for Health in Aging. It provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards. We selected the home safety guide to account for the attention given to the intervention group but not to provide information that would bias the control group away from talking about mammography with the patient's PCP.
  Home safety guide: The home safety guide provides tips about important actions older adults can take to prevent falls, poisoning, and bathroom hazards and protection against abuse, fire and other related hazards.
Arm/Group | Mammogram Decision Aid - Patient | Mammogram Decision Aid - Caregiver | Home Safety Guide - Patient | Home Safety Guide - Caregiver
All-Cause Mortality (participants affected / at risk) | 37/213 | 0/213 | 30/214 | 3/214
Serious Adverse Events (participants affected / at risk) | 1/213 | 0/0 | 2/214 | 0/0
Other Adverse Events (participants affected / at risk) | 4/213 | 0/0 | 4/214 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mammogram Decision Aid - Patient (N=213) | Mammogram Decision Aid - Caregiver (N=0) | Home Safety Guide - Patient (N=214) | Home Safety Guide - Caregiver (N=0)
New Breast Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mammogram Decision Aid - Patient (N=213) | Mammogram Decision Aid - Caregiver (N=0) | Home Safety Guide - Patient (N=214) | Home Safety Guide - Caregiver (N=0)
Complications and distress of receiving a mammogram (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | NA | 4 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03282097/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03282097/ICF_000.pdf